CLINICAL TRIAL: NCT05558280
Title: Maintenance Therapy With Qarziba for Patients in Relapsed/Refractory High-grade Osteosarcoma After Induction Multimodal Therapy - a Phase II Multi-center Study
Brief Title: Qarziba for Patients in Relapsed/Refractory High-grade Osteosarcoma
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: study not started
Sponsor: Prof. Franca Fagioli (Other)
Responsible Party: Sponsor-Investigator, Prof. Franca Fagioli, Professor, Azienda Ospedaliera Ospedale Infantile Regina Margherita Sant'Anna
Organization: Azienda Ospedaliera Ospedale Infantile Regina Margherita Sant'Anna (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MaQ Study
Record Dates: First submitted 2022-09-23; First posted 2022-09-28 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Osteosarcoma in Children
MeSH Terms: interventions — dinutuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dinutuximab beta (Experimental): The treatment phase foresees 5 cycles of Dinutuximab Beta. Dinutuximab Beta administration is restricted to hospital-use only and must be administered under the supervision of a physician experienced in the use of oncological therapies. It must be administered by a healthcare professional prepared to manage severe allergic reactions including anaphylaxis in an environment where full resuscitation services are immediately available. The study treatment will be administered with a continuous intravenous infusion at a dose of 14 mg/mq/day, days 1-5, a total of 60 hours (cumulative dose/cycle: 70 mg/mq). Each cycle lasts 28 days.
  Interventions: Drug: Dinutuximab beta

INTERVENTIONS:
Drug: Dinutuximab beta — The study treatment will be administered with a continuous intravenous infusion at a dose of 14 mg/mq/day, days 1-5, a total of 60 hours (cumulative dose/cycle: 70 mg/mq). Each cycle lasts 28 days.The treatment phase foresees 5 cycles of Dinutuximab Beta.
  Other Names: QARZIBA

SUMMARY:
Limited progress has been made in identifying novel targets that may be therapeutic for Osteosarcoma(OS) and there remains an urgent need for the development of new agents that are effective in improving survival. From this perspective, repurposing already proven targets in other tumors may offer new opportunities for OS in children and young adults. Anecdotal evidence of anti-GD2 therapy exists in OS from prior Phase 1 trials that included patients with OS.

DETAILED DESCRIPTION:
Anecdotal evidence of anti-GD2 therapy exists in OS from prior Phase 1 trials that included patients with OS. In a Phase 1/1B trial of the murine antibody (14.2G2a) plus IL2, 2/33 patients had OS. One patient had multiple bone metastases and received 1 cycle of therapy. Two months later, repeat scans showed a complete response. This patient remained disease free for 8 months but subsequently relapsed.

The Children's oncology group recently investigated the use of dinutuximab monotherapy in patients with recurrent pulmonary OS in complete surgical remission in a single-arm phase II study (AOST1421). Patients received 5 cycles of dinutuximab 70mg/m2/cycle with GM-CSF in 2 different dinutuximab infusion schedules: 35mg/m2/day over 20 hours (2-day) and 17.5mg/m2/day over 10 hours (4-day) schedule. The primary end point was Disease Control Rate (DCR), defined as the proportion of patients' event-free at 12 months from enrollment and success was defined as ≥16/ 39 patients (> 40%) event-free at 12 months from enrollment. The preliminary results of this study were showed at ASCO 2020. Thirty-nine patients were eligible and evaluable (median age 15 yr). One of 136 administered therapy cycles met the criteria for unacceptable toxicity when 1 patient receiving the 2-day schedule died after cycle 2 due to an unknown cause and 1 patient experienced grade 4 neurotoxicity (depressed level of consciousness and respiratory depression) attributed as probably related to the protocol therapy. The protocol was revised to allow only the 4-day schedule. Other ≥ Grade 3 toxicities occurring in > 10 % of participants were predictable dinutuximab toxicities such as pain, diarrhea, hypoxia and hypotension. A DCR of 30.7% (95% CI 17- 47%) was found, as 27/39 patients experienced an event. The final official results have not been published yet, and analyses are ongoing. A humanized version of the anti-GD2 antibody, Naxitamab (hu3F8), developed at Memorial Sloan Kettering Cancer Center, is currently being tested for efficacy against recurrent OS (NCT02502786).

Rationale dose and schedule of Dinutuximab beta in MaQ trial.

The recommended dosage of Dinutuximab (Unituxin, United Therapeutics) is 17.5 mg/m2/day administered IV over 10-20 hours for 4 consecutive days for a maximum of 5 cycles. In AOST1421, patients with recurrent pulmonary OS received 5 cycles of dinutuximab 70mg/m2/cycle with GM-CSF in 2 different infusion schedules: 35mg/m2/day over 20 hours (2-day) (experimental infusion) and 17.5mg/m2/day over 10 hours (4-day) schedule. However, during this trial, 2 serious adverse events (n=1 death, n=1 grade 4 neurotoxicity), possibly related to the experimental infusion schedule of dinutuximab were reported. In light of these events, the protocol was modified for the remainder of the study to allow only the 4-day schedule.

In the EU, Dinutuximab beta is approved for high-risk NB patients at the recommended dosage of 100 mg/m2 per course as either an 8-hour short-term i.v. infusion over 5 consecutive days (STI), or as a long-term i.v. infusion over 10 consecutive days (LTI). A pharmacokinetics study of LTI dinutuximab beta showed that this regimen results in higher plasma exposure at time points preceding subsequent antibody infusions after cycle 1, allowing for a persistent activation of antibody effector mechanisms over the entire treatment period. Moreover, LTI led to a less toxic profile compared with STI regimen. Data on Dinutuximab dosage and safety are based on studies enrolling primary refractory or relapsed NB or first-line NB children with either complete response or at MRD. OS is the most common primary malignant bone tumor in AYA, thus we expect to include older patients than NB patients, that notably experience greater toxicity from antitumor therapies. Moreover, the present trial will enroll patients who have experienced OS R/R and have already received at least one line of standard treatment. Furthermore, so far, PK data are lacking for the adolescent population. For these reasons, the patients enrolled in this study with OS R/R will received Dinutuximab beta (Qarziba) 14 mg/mq/day, for 5 days (total dose: 70mg/sqm/cycle) i.v. continuous infusion. Each cycle will last 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated, written informed consent from each patient or patient's legally acceptable representative, parent (s) or legal guardian in accordance with regional laws or regulations and the patient's assent, when applicable, before any study-specific activity, including screening evaluation, is performed. For patients who reach the age of legal consent during the clinical study, notification may be required and a new consent form may need to be signed by the patient.
* Histologically confirmed high-grade osteosarcoma which is relapsed or refractory (ONLY patients in first or second relapse will be eligible). Histological confirmation from initial diagnosis or relapse is acceptable.
* Disease status: subjects must have achieved a complete or partial response after a second or further line of systemic therapy (with or without surgery) as defined by the following criteria:
* Complete Response = disappearance of all target and non-target lesions
* Partial Response = at least 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD of the last episode of relapse or recurrence. If a partial response is achieved, only patients with a focal localized disease at any site must be enrolled (for patients with lung disease a maximum of 2 lung unilateral nodules will be accepted).
* Age: ≥ 1 to < 25 years old at the time of signing the informed consent form.
* Performance Level: Karnofsky Performance Status ≥ 60% for participants > 16 years old or Lansky Play Score ≥ 60% for pediatric participants ≤ 16 years old. Subjects who are unable to walk because of paralysis and/or previous surgeries will be considered ambulatory for the purpose of assessing their performance score.
* Subjects must have recovered to < Grade 2 per the NCI CTCAE v 4.03 or to baseline from any non-hematologic toxicities (except alopecia) due to previous therapy.
* Life expectancy ≥ 3 months.
* Completed previous line of treatment (systemic therapy with or without surgery) within 28 days prior the first dose of Dinutuximab Beta.
* Adequate bone marrow function independent of transfusion for at least 7 days prior to screening and independent of growth factor support for at least 14 days prior to screening
* Adequate organ function
* Normal ventricular ejection fraction (LV ejection fraction > 50%).
* Availability of paraffin tumor material and/or fresh frozen tumor sample of the most recent biopsy.

Exclusion Criteria:

* Any other malignancy that required treatment within 2 years prior to study drug administration;
* Concomitant Medications:

  * Anticancer agents: subjects who are currently receiving other anticancer agents
  * Corticosteroid: Due to their immunosuppressive activity, concomitant treatment with corticosteroids is not recommend within 2 weeks prior to the first treatment course until 1 week after the last treatment course with Dinutuximab Beta, except for life-threatening conditions
* Prior Therapies and/or Procedures:

  * Major surgery within 28 days prior to the first dose of Dinutuximab Beta.
  * Minor surgery within 14 days prior to the first dose of Dinutuximab Beta.
  * Received prior to treatment with Dinutuximab Beta or any other monoclonal antibody GD2.
  * Received prior to treatment with chimeric antigen receptor anti GD2 therapy (CAR-T anti GD2) within 28 days prior to the first dose of Dinutuximab Beta.
  * Received any anti-cancer drug within 28 days prior to the first dose of Dinutuximab Beta.
  * Received any investigational drug within 28 days prior to the first dose of Dinutuximab Beta.
  * Received radiotherapy or proton-therapy within 28 days prior to the first dose of Dinutuximab Beta.
  * Received any immunotherapy within 28 days prior to the first dose of Dinutuximab Beta.
  * Received any live (including attenuated) vaccines within 28 days prior the first dose of Dinutuximab Beta.
* Disease progression or presence of a multifocal disease after the induction therapy (except for the presence of only 2 unilateral lung diseases).
* Has hypersensitivity to either study drug or any of the excipients.
* Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, cardiac arrhythmia, auto-immune disease or psychiatric illness or social situations that would limit compliance with study requirements, substantially increase risk of incurring AEs from IP.
* Active infection including hepatitis B (known positive hepatitis B virus [HBV] surface antigen [HbsAg]), hepatitis C, HIV (positive HIV 1/2 antibodies). Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody and absence of HbsAg) are eligible. Patients positive for hepatitis C virus (HCV) antibody are eligible only if the polymerase chain reaction is negative for HCV ribonucleic acid (RNA).
* Has peripheral or central neuropathy ≥ Grade 2 (CTCAE v 4.03).
* Has photophobia ≥ Grade 2 (CTCAE v 4.03).
* Has uncontrolled seizure disorder.
* Females who are pregnant or lactating.
* Willingness to avoid pregnancy or fathering children

Ages: 1 Year to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 22 (Estimated)
Dates: Start 2023-11-30 (Estimated); Primary Completion 2025-12-15 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
Efficacy of Dinutuximab Beta as maintenance therapy in patients with OS relapsed/refractory that have achieved Complete Response (CR) or Partial Response (PR) | 12months
  • Disease Control Rate (DCR) at 12 months from the last episode of relapse/refractory patients with CR or PR OS R/R treated with a maintenance therapy with Dinutuximab Beta.

CONTACTS AND LOCATIONS:
Overall Officials: Franca Fagioli, MD, Principal Investigator — A.O.U. Città della Salute e della Scienza
Locations (1):
- AOU Città della Salute e della Scienza di Torino - Presidio Infantile Regina Margherita, Turin, Italy

IPD SHARING:
Plan to Share IPD: No